CLINICAL TRIAL: NCT00645814
Title: Multicenter Study of the Safety and Efficacy of Adalimumab in Subjects With Moderate to Severe Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Beverly Paperiello / Director, Clinical Program Management, Abbott
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M02-528
Record Dates: First submitted 2008-03-26; First posted 2008-03-28 (Estimated); Last update posted 2008-03-28 (Estimated); Status verified 2008-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Placebo Comparator)
  Interventions: Drug: placebo for adalimumab
- B (Active Comparator)
  Interventions: Drug: adalimumab
- C (Active Comparator)
  Interventions: Drug: adalimumab

INTERVENTIONS:
Drug: placebo for adalimumab — 80 mg at Week 0 and 40 mg eow through Week 11
  Other Names: placebo
  Arms: A
Drug: adalimumab — 80 mg at Week 0 and 40 mg eow through Week 11
  Other Names: ABT-D2E7; Humira
  Arms: B
Drug: adalimumab — 80 mg at Week 0 and 40 mg weekly through Week 11
  Other Names: ABT-D2E7; Humira
  Arms: C

SUMMARY:
Study of the Safety and Efficacy of Adalimumab in Subjects with Moderate to Severe Chronic Plaque Psoriasis

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate to severe chronic plaque psoriasis
* Active psoriasis, despite topical therapies

Exclusion Criteria:

* Other active skin diseases or skin infections
* Prior exposure to any anti-TNF therapy
* Subject has other active skin diseases
* Multiple concomitant therapy restrictions and/or washouts (topicals, UV, other systemic PS therapies)
* Poorly controlled medical conditions
* History of neurologic symptoms suggestive of central nervous system (CNS) demyelinating disease.
* History of cancer or lymphoproliferative disease
* History of active TB or listeriosis, or persistent chronic or active infections
* Known to have immune deficiency or is immunocompromised
* Clinically significant abnormal laboratory test results
* Erythrodermic psoriasis or generalized pustular psoriasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2003-03; Primary Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Psoriasis Area and Severity Index | Week 12
Adverse Events | Throughout Study Participation

SECONDARY OUTCOMES:
Psoriasis Area and Severity Index | Week 1, 2, 4, 8, 12
DLQI, SF-36, Zung Depression Self-Rating Scale, EQ-5D | Week 12

REFERENCES:
- [Derived] Ryan C, Sobell JM, Leonardi CL, Lynde CW, Karunaratne M, Valdecantos WC, Hendrickson BA. Safety of Adalimumab Dosed Every Week and Every Other Week: Focus on Patients with Hidradenitis Suppurativa or Psoriasis. Am J Clin Dermatol. 2018 Jun;19(3):437-447. doi: 10.1007/s40257-017-0341-6. PMID 29380251
- [Derived] Papp KA, Armstrong AW, Reich K, Karunaratne M, Valdecantos W. Adalimumab Efficacy in Patients with Psoriasis Who Received or Did Not Respond to Prior Systemic Therapy: A Pooled Post Hoc Analysis of Results from Three Double-Blind, Placebo-Controlled Clinical Trials. Am J Clin Dermatol. 2016 Feb;17(1):79-86. doi: 10.1007/s40257-015-0161-5. PMID 26547918